CLINICAL TRIAL: NCT04257682
Title: Comparing Efficacy and Safety of Three Regional Anesthesia Regimens in Total Hip and Knee Arthroplasty: A Double Blind Randomized Control Trial
Brief Title: Regional Anesthesia in Total Hip and Knee Arthroplasty
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20190297-01H
Record Dates: First submitted 2019-12-20; First posted 2020-02-06 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2022-08

CONDITIONS: Knee Osteoarthritis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Bupivacaine; Anesthetics, Local; Ropivacaine; Mepivacaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bupivacaine (Active Comparator): The participant will receive Bupivacaine as anesthesia during his or her planned total hip or knee replacement surgery.
  Interventions: Drug: Bupivacaine
- Ropivacaine (Active Comparator): The participant will receive Ropivacaine as anesthesia during his or her planned total hip or knee replacement surgery.
  Interventions: Drug: Ropivacaine
- Mepivacaine (Active Comparator): The participant will receive Mepivacaine as anesthesia during his or her planned total hip or knee replacement surgery.
  Interventions: Drug: Mepivacaine

INTERVENTIONS:
Drug: Bupivacaine — Bupivacaine is a long-lasting dense sensory-motor block that can last up to four hours. It will be administered once, as part of the spinal anesthetic. The dosage varies based on age and joint, from 6.75 mg to 8.25 mg for the knee, and 7.5 mg to 9 mg for the hip.
  Other Names: Local Anesthetic
  Arms: Bupivacaine
Drug: Ropivacaine — Ropivacaine is a long-acting local anesthetic that is known for its differential sensory-motor block. It will be administered once, as part of the spinal anesthetic. The dosage varies based on age and joint, from 9 mg to 11 mg for the knee, and 10 mg to 12 mg for the hip.
  Other Names: Local Anesthetic
  Arms: Ropivacaine
Drug: Mepivacaine — Mepivacaine is an intermediate-acting local anesthetic producing shorting and motor-sparing blocks. It will be administered once, as part of the spinal anesthetic. The dosage varies based on age and joint, from 40 mg to 50 mg for the knee, and 45 mg to 55 mg for the hip.
  Other Names: Local Anesthetic
  Arms: Mepivacaine

SUMMARY:
The purpose of this study is to test whether the use of Ropivacaine and Mepivacaine are better in terms of effectiveness, cost, and safety than Bupivacaine as regional anesthetics in elective hip or knee replacement surgery.

DETAILED DESCRIPTION:
Advances in pain management, regional anesthesia, and focused rehabilitation have increased the popularity of outpatient total hip and knee arthroplasty in a select group of eligible patients. However, one of the main impediments to same-day discharge is the prolonged motor block post-spinal anesthesia, as patients are routinely kept in the post-anesthesia care unit (PACU) until they demonstrate that the spinal anesthesia has worn off.

At The Ottawa Hospital, the standard treatment for people receiving anesthesia during a total arthroplasty is the use of the anaesthetic, Bupivacaine. Mepivacaine and Ropivacaine are alternative anaesthetics that are also in use at The Ottawa Hospital. They are growing in popularity as anaesthetics because they and allow quicker recovery time when compared to Bupivacaine. Bupivacaine results in a long-lasting sensory-motor block, meaning that in the area that the local anesthesia was used, there is no sensation and limited movement for long periods of time. During hip or knee replacement surgery, you may want to have no sensation and the inability to move your lower limbs. However, it is not ideal for after surgery where weakness in the legs puts a person at increased risk for falls. Therefore, hospitalization after surgery typically lasts for a longer duration. Mepivacaine and Ropivacaine have a shorter motor block duration, allowing for a potentially earlier hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total hip or knee replacement

Exclusion Criteria:

* Study refusal
* Inability to provide consent
* Contra-indications to spinal anesthesia (refusal, infection, anti-coagulation, bleeding diathesis)
* Bilateral surgery
* Revision surgery
* Pre-exiting chronic pain or opioid consumption ≥ 30mg oxycodone or equivalent
* Pregnancy
* Not receiving preoperative adductor canal block for any reason
* Contra-indication to multimodal analgesia (acetaminophen or NSAIDs)
* Obstructive sleep apnea requiring extended PACU stay
* History of severe postoperative nausea and vomiting

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Compare the effectiveness of Ropivacaine and Mepivacaine spinal anesthetics to the current standard of care using Bupivacaine: proportion of patients with a failed spinal anesthetic | Day of surgery
  Effectiveness will be measured by looking at the proportion of patients with a failed spinal anesthetic.
Compare the cost profile of Ropivacaine and Mepivacaine spinal anesthetics to the current standard of care using Bupivacaine. | Hospital discharge, approximately 1 day
  Total costs associated with the providers involved and the costs associated with the time spent in the hospital following surgery but before discharge will be combined to report the cost profile

SECONDARY OUTCOMES:
Compare changes in post-operative pain associated with Ropivacaine and Mepivacaine spinal anesthetics to the current standard of care using Bupivacaine. | Immediately after completion of surgery, every hour during PACU stay - approximately 3 hours, every 6 hours during hospital stay - approximately 1 day, 24 hours after surgery, one week post-operatively
  Post-operative pain will be measured using a combination of the Visual Analogue Scale Pain Scores (VAS), time to first analgesic request in PACU, and recording post-operative opioid use.
Compare the safety of Ropivacaine and Mepivacaine spinal anesthetics to the current standard of care using Bupivacaine. | 24 hours after surgery, one week post-operatively
  Safety parameters will be compared by recording Adverse Events (AE)
Compare the quality of the block provided by Ropivacaine and Mepivacaine spinal anesthetics to the current standard of care using Bupivacaine. | During surgery, PACU discharge - approximately 3 hours
  Quality of the block will compared by combing the the duration of total sensory and motor blocks and the number of patients who do not achieve a block at time of incision.
Compare the length of stay for patients who received Ropivacaine and Mepivacaine spinal anesthetics to the current standard of care using Bupivacaine. | Immediately after surgery, PACU discharge - approximately 3 hours, SDC discharge - approximately 1 day, hospital discharge - approximately 1 day
  Length of stay will be compared by recording the time of PACU discharge, SDC discharge, and hospital discharge.